CLINICAL TRIAL: NCT03762096
Title: Short Interval Resveratrol Trial in Cardiovascular Surgery
Acronym: SIRT-CVS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Douglas B. Sawyer, Chief Academic Officer, MaineHealth
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1095584
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resveratrol (Experimental)
  Interventions: Dietary Supplement: Trans-resveratrol
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Trans-resveratrol — 1 gram, twice a day by mouth Transmax (Biotivia)
  Other Names: resveratrol
  Arms: Resveratrol
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Major Problem

People with diabetes have an increased risk of heart disease, heart failure, and death from a cardiovascular cause. Diabetes prevents efficient metabolism of fuel, causes inflammation and vascular disease that blocks normal blood flow, and inhibits the function of the heart after injury. These changes make diabetics more susceptible to heart attacks and heart failure.

Resveratrol is found in grapes and red wine and has been shown to have beneficial effects in diabetic patients. In previous studies the investigators have shown that resveratrol can improve heart metabolism and function in pigs with diabetes and chronic lack of blood flow to the heart.

Questions

The investigators believe resveratrol will help reverse the negative effects of diabetes on the heart. The questions are: 1.How does the molecular machinery in the hearts of patients with diabetes differ from patients without diabetes? 2.Will resveratrol have an effect on heart metabolism, intracellular signaling, inflammation and blood vessel function? 3.Will resveratrol improve the number and function of cardiac stem cells, cells involved in heart repair? The investigators have been safely collecting tissue from the hearts of patients undergoing heart surgery. Preliminary studies show the investigators can isolate and study cells. The investigators have collected and assessed the function of endothelial cells, a measure of vascular health and can measure the level of endothelial injury and have studied the make-up of caveolae, structures on the cell membrane that are important for cell signaling and are negatively impacted by diabetes. This study is a unique collaboration among cardiologists, cardiac surgeons, and basic scientists.

DETAILED DESCRIPTION:
Patients with diabetes and metabolic diseases such as obesity, hypertension and dyslipidemia have a myocardial environment that results in endothelial dysfunction, altered metabolism and little potential for regeneration by intrinsic or extrinsically delivered therapies. Based upon work in animal and cell culture models of human disease, caveolae, lipid rafts found on the cell membrane of endothelial cells and myocytes, are important in cell signaling and metabolism. A growing body of literature suggests that disruption of membrane lipid microdomains in diabetes can lead to altered signaling that contributes to cardiovascular pathology. One possible method to improve the "endothelial health" of the heart could involve normalizing metabolic processes and decreasing signals that lead to inflammation and pathways that lead to fibrosis in the myocardium. This presents an opportunity to improve outcomes in our diabetic patients and improve the success of future therapies aimed at improving endothelial function.

Resveratrol, a polyphenol found in abundance in red wine, activates sirtuin 1 (SIRT1), an NAD+-dependent deacetylase, which influences a diverse array of metabolic pathways. Studies in cultured cells, small animal models, and humans demonstrate that SIRT1 is involved in endothelial function, mitochondrial biogenesis, insulin production, inflammation, and glucose and lipid homeostasis. These processes are often dysfunctional in patients with diabetes and other metabolic diseases.

The central hypothesis of this proposal is that molecular pathology of diabetes on cardiac endothelium can be corrected with orally supplemented resveratrol.

The investigators propose to test this hypothesis in by first assessing endothelial function, lipidomic signatures, and cell signaling in patients with and without diabetes mellitus undergoing coronary artery bypass grafting (CABG) with cardiopulmonary bypass (CPB). The second Aim of this proposal is a pilot placebo-controlled, double-blind clinical trial that will assess the effects of supplemental resveratrol in diabetic patients undergoing CABG with CPB. The goal will be to better understand the influence of resveratrol on key molecular signals that determine endothelial function, calveolar makeup and function, as well as cytoprotective signaling and responses in the heart.

The Specific Aims of this proposal are to:

Aim 1: Define the molecular pathology of diabetes on cardiac cells and tissues in non-diabetic and diabetic patients undergoing surgical revascularization. We will assess the effects of DM on endothelial function and damage, lipidomics, caveolar expression, disrupted receptor expression and neuregulin signaling.

Aim 2: Determine the effect of resveratrol on the microvascular function of diabetic patients undergoing surgical revascularization. Through a pilot randomized placebo-controlled clinical trial, the investigators will evaluate the effect of resveratrol on endothelial damage at the time of cardiopulmonary bypass, endothelial function, and cell signaling.

This study will further our understanding of how resveratrol impacts patients in a controlled setting, and will allow for a thorough and complete investigation of how the supplement affects this patient population clinically and on a molecular level. The data will inform the development of larger studies examining the benefits of resveratrol in diabetes and metabolic syndrome. Finally, the investigators successful completion of this trial will inform the study of other therapeutics where direct myocardial effects are being considered.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18 years)
* Type 2 diabetes (controlled by either oral agents or insulin)
* Coronary artery disease referred for elective CABG with CPB

Exclusion Criteria:

* Known decompensated congestive heart failure or systolic heart failure with an ejection fraction < 45% at the time of evaluation
* Liver Function Tests (LFT) greater than 2 times normal
* Renal dysfunction (GFR less than 60 mL/min)
* Abnormal coagulation profile (PT/PTT and INR)
* Alcohol consumption more than 3 grams (equivalent to 2.5 glasses of wine) daily
* Positive HIV, Hepatitis B or C testing
* Severe ventricular arrhythmias
* Significant hypotension (SBP < 90 mmHg) at the time of enrollment
* Patients who are pregnant
* Known malignancy other than non-melanoma skin cancers
* Expected survival less than one year.
* Allergy or intolerance to the ingredients of the supplement or the placebo
* Inability to comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-06 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in endothelial function | 6 weeks
  Serum levels of nitric oxide (ELISA assay)
Change in endothelial function | 14 days
  Nitric oxide synthase levels in heart tissue (Western blot assay)

SECONDARY OUTCOMES:
Effects of resveratrol on caveolar function | 14 days
  Lipidomic changes in cell membranes (Mass spectrometry)
Effects of resveratrol on molecular signaling | 14 days
  Serum and tissue levels of pathways associated with glucose metabolism (Western blot assay)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Sawyer, Principal Investigator — Maine Health
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No